CLINICAL TRIAL: NCT00180817
Title: Longitudinal Study of the Clinical and Haematological Cause of Women With Antiphospholipid Antibodies in Women Presenting as Recurrent Miscarriages.
Brief Title: Longitudinal Study of the Clinical and Haematological Cause of Women With Antiphospholipid Antibodies.
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: EC3103
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Antiphospholipid Syndrome
Keywords: Antiphospholipid syndrome
MeSH Terms: conditions — Antiphospholipid Syndrome

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
This study is being done to see if there are any long term health related issues in women with APA and recurrent miscarriages.

DETAILED DESCRIPTION:
The association between APA and thrombosis is well documented. Both LA and ACA are often detected in individuals with SLE but there is no prospective data on the risk of thrombosis in women who present with recurrent miscarriages in association with APA. This study should significantly advance medical knowledge of the natural history of primary antiphospholipid syndrome (PAPS) which is essential to enable optimal management of relatively young women who may be at risk of complications, some of which are potentially life threatening.

ELIGIBILITY:
Inclusion Criteria:

Antiphospholipid syndrome History of recurrent miscarriages

Exclusion Criteria:

Previous thromboembolic disease

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 1998-09 (Actual); Primary Completion 2005-08-31 (Actual); Study Completion 2005-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lesley Regan, Principal Investigator — Imperial College London; Raj Rai, MRCOG, Principal Investigator — Imperial College London; Winnie Lo, Principal Investigator — St. Mary's NHS Trust, London; Preeti Jindal, MRCOG, Principal Investigator — St. Mary's NHS Trust, London
Locations (1):
- St. Mary's Hospital, London, United Kingdom